CLINICAL TRIAL: NCT00394459
Title: Randomised, Prospective, Single-blind, Controlled Multicenter Study on the Safety of Two Epidural Catheters in Patients Undergoing Surgery Under Thoracic Epidural Anaesthesia
Brief Title: Safety of Two Epidural Catheters in Thoracic Epidural Anaesthesia (TEA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Marco Marcus, MaastrichtUMC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC 04-1-83; H-04-078-04
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Anesthesia, Epidural; Paraesthesia
Keywords: Anaesthetic techniques; epidural; catheters; paraesthesia; side effects; Anesthesia, Epidural [E03.155.086.131]
MeSH Terms: conditions — Paresthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Perifix Standard
  Interventions: Device: Perifix Epidural Anaesthesia Catheter; Device: Perifix Standard
- B (Experimental): Perifix New
  Interventions: Device: Perifix Epidural Anaesthesia Catheter; Device: Perifix New

INTERVENTIONS:
Device: Perifix Epidural Anaesthesia Catheter — Epidural Catheter
Device: Perifix Standard — Perifix Standard
  Arms: A
Device: Perifix New — Perifix New
  Arms: B

SUMMARY:
Primary Objective: The primary objective is to demonstrate that the safety of Perifix New is non-inferior to using Perifix Standard when applied for thoracic epidural anaesthesia.

Primary Endpoint: Incidence of spontaneous paraesthesia during catheter insertion

Secondary Objectives: The secondary objectives are to determine the safety and performance of the investigational product: frequency of inadvertent vascular cannulation, difficulties involved in insertion and removal of the catheter, other safety features and data for the evaluation of handling characteristics.

Title: Randomised, prospective, single-blind, controlled, study on the safety of two epidural catheters in patients undergoing surgery under thoracic epidural anaesthesia

Investigational Product: Perifix Epidural Anaesthesia Catheter

Test Product: Perifix New

Reference Product: Perifix Standard

Number of Sites and Countries: 1 site in The Netherlands

Indication: Thoracic epidural anaesthesia

Study Design: Randomised, prospective, single-blind, controlled study in 1 study center, phase IV

Perifix New and Perifix Standard meet all the appropriate provisions of the relevant legislation implementing European Directives (both have CE-marking).

Study Duration: 2 year duration

Study Start: March-April 2005

Sample Size: n = 2*70 patients

DETAILED DESCRIPTION:
Epidural anaesthesia is a central neuraxial block technique with many applications. Improvements in equipment, drugs and technique have made it a popular and versatile anaesthetic technique, with applications in surgery, obstetrics and pain control. Both single injection and catheter techniques can be used. Its versatility means it can be used as an anaesthetic, as an analgesic adjuvant to general anaesthesia, and for postoperative analgesia in procedures involving the lower limbs, perineum, pelvis, abdomen and thorax.

Although epidural anaesthesia is a safe technique, during the insertion of epidural catheters several side effects may occur, including transient paraesthesia and inadvertent vascular cannulation.

Reported incidences for paraesthesia vary widely between about 0.2% and 50% in different articles, depending on the catheter (catheter material, soft-tipped or firm-tipped catheter), the applied technique (lumbar or thoracic epidural anaesthesia, depth of catheter insertion), the approach (midline or paramedian) and the included patients (obstetrical or non-obstetrical). Paraesthesias are not supposed to lead to permanent neurological sequelae, but are unpleasant and perturbing sensations for the patient.

Besides inadvertent intrathecal location of the catheter, further problems include technical difficulties during threading or removal of the catheter. Here, the catheter shaft material seems to be the crucial factor for the incidence of problems.

Based upon years of experience, a wide range of epidural catheters were created, among them the Perifix catheter of B. Braun. Common features are their high tensile strength and stretch resistance, excellent shaft stability with easy visualisation of blood or spinal fluid due to the crystal clear material, no risk of forming loops or knots, and softening of catheter within a few hours due to water absorption of the polyamide material.

Recently, B. Braun Melsungen AG has developed a new generation of Perifix epidural catheters, which are already CE-labeled. These new catheters are different in their composition compared to the current Perifix Standard catheter with regard to the catheter material and tip configuration. They have an outer poly-urethane liner and an inner polyamide body. Experimental tests have shown that the positive features (e.g. pushability, kink resistance, gliding, withdrawal) of the Perifix Standard catheter can be maintained. Due to the polyurethane outer layer, the catheter gets softer when reaching body temperature immediately upon insertion. Based on this, it is expected that paraesthesias during catheter injection can be reduced by at least 20%.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thoracic epidural anaesthesia (TEA), with or without general anaesthesia.
* American Society of Anesthesiologists (ASA) class I-III
* Patients aged 18 and ≤ 75 years of age

Exclusion Criteria:

* Anamnestic exclusion criteria are all contraindications for epidural anaesthesia.
* Severe scoliosis, previous surgery on the spine, M. Bechterew disease
* Non-competent and non-cooperative patients
* Patients with medicament and drug abuse problems, problems in communication, participating in parallel in another clinical study with experimental drugs or devices, receiving prohibited concomitant therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-04; Primary Completion 2008-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary end-point will be the incidence of spontaneous paraesthesia during catheter insertion in TEA-patients. | 1 hour

SECONDARY OUTCOMES:
The frequency of inadvertent vascular cannulation | 1 hour
Difficulties involved in insertion and removal of the catheter | 1 week
Data on additional complications | 1 week
Data for the evaluation of handling characteristics | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Gielen, MD, PhD, Study Chair — Radboud University Medical Center; Marco Marcus, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands